CLINICAL TRIAL: NCT06680011
Title: Cohort-Based Study of Diagnostic Biomarkers for Neurosyphilis
Status: Recruiting | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Other Study IDs: smhcgxy_2
Record Dates: First submitted 2024-10-23; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-10

CONDITIONS: Neurosyphilis; Biomarkers; Proteomics
MeSH Terms: conditions — Neurosyphilis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, cerebrospinal fluid, and stool samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Neurosyphilis Patients: 1. Meet the diagnostic criteria for neurosyphilis in this study based on the 2015 Sexually Transmitted Diseases Treatment Guidelines published by the Centers for Disease Control and Prevention (CDC) and the 2020 European Guideline on the Management of Syphilis: ① Positive serological tests for Treponema pallidum (e.g., Treponemal tests) and rapid plasma reagin (RPR) tests; ② Positive cerebrospinal fluid tests for Treponema pallidum particle agglutination assay (TPPA), the toluidine red unheated serum test (TRUST), and the Venereal Disease Research Laboratory test (VDRL).
  2. Aged 18-65 years, regardless of gender (female patients are rare in clinical practice).
  3. At least a junior high school education level, with sufficient auditory and visual function to complete the necessary examinations and assessments for this study.
  4. No contraindications for electroencephalogram (EEG) and transcranial magnetic stimulation (TMS).
- Non-neurosyphilis Syphilis Patients: 1. Positive serological tests for Treponema pallidum (e.g., Treponemal tests) and rapid plasma reagin (RPR) tests.
  2. Does not meet the diagnostic criteria for neurosyphilis in this study, based on the 2015 Sexually Transmitted Diseases Treatment Guidelines published by the Centers for Disease Control and Prevention (CDC) and the 2020 European Guideline on the Management of Syphilis: ① Positive serological tests for Treponema pallidum and rapid plasma reagin tests; ② Positive cerebrospinal fluid tests for Treponema pallidum particle agglutination assay (TPPA), the toluidine red unheated serum test (TRUST), and the Venereal Disease Research Laboratory test (VDRL).
  3. Aged 18-65 years, regardless of gender (female patients are rare in clinical practice).
  4. At least a junior high school education level, with sufficient auditory and visual function to complete the necessary examinations and assessments for this study.
  5. No contraindications for electroencephalogram (EEG).
- Healthy Controls: 1. Physically healthy (no mental illnesses or diseases affecting bodily organs).
  2. Aged 18-65 years, regardless of gender.
  3. At least a junior high school education level, with sufficient auditory and visual function to complete the necessary examinations and assessments for this study.
  4. No contraindications for electroencephalogram (EEG).

SUMMARY:
The goal of this observational study is to identify diagnostic biomarkers for neurosyphilis in patients with the condition. The main questions it aims to answer are:

What plasma biomarkers are associated with neurosyphilis? What electrophysiological characteristics (EEG and eye movement) are linked to neurosyphilis? Researchers will compare biomarker data from plasma and gut microbiome analyses with electrophysiological findings to see if these factors can help diagnose neurosyphilis.

Participants will:

Provide clinical information such as age, gender, symptoms, and disease course Submit blood and urine samples for proteomics and metagenomic sequencing Undergo EEG and eye movement evaluations for electrophysiological analysis

ELIGIBILITY:
Inclusion Criteria:

* Neurosyphilis Patients

  1. Meet the diagnostic criteria for neurosyphilis in this study based on the 2015 Sexually Transmitted Diseases Treatment Guidelines published by the Centers for Disease Control and Prevention (CDC) and the 2020 European Guideline on the Management of Syphilis: ① Positive serological tests for Treponema pallidum (e.g., Treponemal tests) and rapid plasma reagin (RPR) tests; ② Positive cerebrospinal fluid tests for Treponema pallidum particle agglutination assay (TPPA), the toluidine red unheated serum test (TRUST), and the Venereal Disease Research Laboratory test (VDRL).
  2. Aged 18-65 years, regardless of gender (female patients are rare in clinical practice).
  3. At least a junior high school education level, with sufficient auditory and visual function to complete the necessary examinations and assessments for this study.
  4. No contraindications for electroencephalogram (EEG) and transcranial magnetic stimulation (TMS).
* Non-neurosyphilis Syphilis Patients

  1. Positive serological tests for Treponema pallidum (e.g., Treponemal tests) and rapid plasma reagin (RPR) tests.
  2. Does not meet the diagnostic criteria for neurosyphilis in this study, based on the 2015 Sexually Transmitted Diseases Treatment Guidelines published by the Centers for Disease Control and Prevention (CDC) and the 2020 European Guideline on the Management of Syphilis: ① Positive serological tests for Treponema pallidum and rapid plasma reagin tests; ② Positive cerebrospinal fluid tests for Treponema pallidum particle agglutination assay (TPPA), the toluidine red unheated serum test (TRUST), and the Venereal Disease Research Laboratory test (VDRL).
  3. Aged 18-65 years, regardless of gender (female patients are rare in clinical practice).
  4. At least a junior high school education level, with sufficient auditory and visual function to complete the necessary examinations and assessments for this study.
  5. No contraindications for electroencephalogram (EEG).
* Healthy Controls

  1. Physically healthy (no mental illnesses or diseases affecting bodily organs).
  2. Aged 18-65 years, regardless of gender.
  3. At least a junior high school education level, with sufficient auditory and visual function to complete the necessary examinations and assessments for this study.
  4. No contraindications for electroencephalogram (EEG).

Exclusion Criteria:

* Neurosyphilis Patients & Non-neurosyphilis Syphilis Patients

  1. Age < 18 years or > 65 years;
  2. Pregnant or breastfeeding women (female patients are rare in clinical practice);
  3. HIV-positive;
  4. Presence of severe primary diseases (such as liver, kidney, endocrine, or hematological diseases) accompanied by autoimmune diseases or connective tissue diseases;
  5. Presence of other central nervous system diseases besides neurosyphilis;
  6. Contraindications for transcranial magnetic stimulation (TMS) treatment, such as history of head trauma, epilepsy, or presence of metal implants;
  7. Contraindications for electroencephalography (EEG), such as severe scalp injuries, extensive or open cranial trauma, inability to place electrodes, or potential for infection from the examination.
  8. Education level below junior high school.
* Healthy Controls

  1. Age < 18 years or > 65 years;
  2. Pregnant or breastfeeding women;
  3. HIV-positive;
  4. Other central nervous system diseases, severe physical illnesses, or major organ diseases;
  5. Presence of severe primary diseases (such as liver, kidney, endocrine, or hematological diseases) accompanied by autoimmune diseases or connective tissue diseases;
  6. Contraindications for electroencephalography (EEG), such as severe scalp injuries, extensive or open cranial trauma, inability to place electrodes, or potential for infection from the examination;
  7. Education level below junior high school.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of neurosyphilis patients, non-neurosyphilis syphilis patients, and healthy controls aged 18-65.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Measurement of AIM2 inflammasome in peripheral blood. | Data will be collected at baseline, 6 months, and 12 months after enrollment.
  This measure will assess the expression levels of the AIM2 inflammasome in peripheral blood samples from subjects using proteomics methods, mass spectrometry.
Measurement of NFL and sTREM2 in cerebrospinal fluid. | Data will be collected at baseline, 6 months, and 12 months after enrollment.
  This measure will evaluate the levels of neurofilament light chain (NFL) and myeloid cells 2 (sTREM2) in cerebrospinal fluid samples from subjects. The measurement will utilize techniques such as TRUST, TPPA and mass spectrometry to assess these biomarkers.

SECONDARY OUTCOMES:
Assessment of Cognitive Function using MoCA | Cognitive assessments will be conducted at baseline and 6 months post-enrollment.
  This measure will evaluate cognitive function in subjects using the Montreal Cognitive Assessment (MoCA).
  The MoCA is a 30-point test that assesses multiple cognitive domains, including visuospatial and executive functions, naming, memory, attention, language, and orientation. Higher scores indicate better cognitive function, with a maximum possible score of 30. A score of 26 or above is considered within the normal range, while a score of 25 or below may indicate mild cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China